CLINICAL TRIAL: NCT04276246
Title: Supplementary Implants Supporting Conventional RDPs in Kennedy Class I: A Dual-centered Randomized Controlled Trial
Brief Title: Supplementary Implants Supporting Conventional Removable Dental Prosthesis (RDPs) in Kennedy Class I
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: ITI International Team for Implantology, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-02167; ex19Joda2
Record Dates: First submitted 2020-02-06; First posted 2020-02-19 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Partial Edentulism Kennedy Class 1
Keywords: Partial Edentulism; Kennedy Class 1; Removable partial dentures (RPDs); Supplementary implants
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): All included participants receive each side 1 posterior implant in the edentulous areas bilaterally in Kennedy class I. Participants are provided with a conventional clasp retained removable partial denture (RPD) worn for 3 months. When implant osseointegration is ensured (3 months healing period), patients are assigned to retentive components (Group A, Test) which are connected to the implants to retain the RPD
  Interventions: Device: dental implants and retentive implant components
- Control (Experimental): All included participants receive each side 1 posterior implant in the edentulous areas bilaterally in Kennedy class I. Participants are provided with a conventional clasp retained removable partial denture (RPD) worn for 3 months. When implant osseointegration is ensured (3 months healing period), patients are assigned to supportive components (Group B, Control), which are connected to the implants to support the RPD
  Interventions: Device: dental implants and supportive implant components

INTERVENTIONS:
Device: dental implants and retentive implant components — retentive components (Group A Test), which are connected to the implants to retain the RPD
  Arms: Experimental
Device: dental implants and supportive implant components — supportive components (Group B Control), which are connected to the implants to support the RPD
  Arms: Control

SUMMARY:
In this study the additional effect of supplementary implants in patients with Kennedy Class I in terms of patient-reported outcome measures (PROMs) and cost-benefit-analyses comparing costs of maintenance care will be investigated

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have voluntarily signed the informed consent before any study action, are willing and able to attend scheduled follow-up visits, and agree that the encoded data will be collected and analyzed
* Males and females with at least 18 years of age
* intraoral situation with bilateral edentulous areas located posterior to the remaining natural teeth (Kennedy class I) in the upper or lower jaw
* remaining dentition includes a first premolar, canine or incisor as the most posterior tooth

Exclusion Criteria:

* Uncontrolled systemic disease that would interfere with dental implant therapy;
* Patients who smoke > 10 cigarettes per day or tobacco equivalents;
* Patients with alcohol and/or drug abuse;
* Patients with chronic pain;
* Patients with untreated periodontitis and / or inadequate oral hygiene (Plaque Index < 30%);
* Medical conditions requiring chronic high dose steroid therapy or anti-resorptive treatment;
* Conditions or circumstances, in the opinion of the investigators, which would prevent completion of study participation or interfere with analysis of study results such as history of non-compliance or unreliability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-02-06 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Changes in patient-reported outcome measures (PROM) | assessment before implant placement, -1 week and 3 months after RPD insertion, 1 week and 3 months after connecting the implant components, 1 to 5 years after implant placement (5-year study period)
  Assessment of patient's perception of function and oral health comparing conventional RPDs to implant-supported RPDs with and without retentive components in posterior sites of Kennedy Class I. PROMs are evaluated using the Oral Health Impact Profile (OHIP 14), i.e. the short form of OHIP with 14 items measuring oral health-related quality of life (OHQoL). The frequency of impairment in different areas (functional limitation, physical discomfort or disability, psychological discomfort or disability, social disability, and handicap) are indicated on a multi-level scale ("never"=0, "hardly"=1, "sometimes"=2, "often"=3, "very often"=4)
Changes in chewing efficiency | assessment before implant placement, -1 week and 3 months after RPD insertion, 1 week and 3 months after connecting the implant components, 1 to 5 years after implant placement (5-year study period)
  Assessment of the chewing Efficiency by masticating standardized fruit gum with three varying degree of hardness. A complete chewing function test comprises 9 chewing sequences: the different hardness of the model food is chewed once on the right, then on the left and finally on both sides. The study participants have 30 seconds for each chewing sequence and 30 seconds between each chewing sequence. Only one fruit gum is chewed per chewing sequence. The samples are placed on a defined area, photographed in standardized manner and analyzed with a computer program. The mean size and amounts of the chewed particles are calculated and determines the chewing efficiency

SECONDARY OUTCOMES:
prosthetic and implant survival rates | during follow-ups, 1 of 5 years after implant placement
  prosthetic and implant survival rates (%) accounting for any technical and biological complication over 5 years
cost-benefit-analyses | during follow-ups, 1 of 5 years after implant placement
  cost-benefit-analyses over time, including costs during maintenance care during follow-up of 5 years will be conducted to compare test and control
Evaluation of success of entire treatment | during follow-ups, 1 of 5 years after implant placement
  evaluation of success of the entire treatment including assessments of technical (prosthesis adjustment or implant abutment adjustment or exchange) and biological complications (peri-implant diseases)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Reconstructive Dentistry, University Center for Dental Medicine Basel UZB, University of Basel, Basel, Switzerland